CLINICAL TRIAL: NCT04067401
Title: Career Enhancement Training Study (USAF)
Acronym: CETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Wyman, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1337
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: The study design will involve randomizing approximately 1440 Airman-in-Training (AiT) within 160 Technical Training classes to one of two conditions: Wingman-Connect or a brief Stress Management training. Randomization will occur at the class level, since Wingman-Connect is designed to train AiTs within a class together as a group (those who voluntarily enroll).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wingman Connect (Experimental): Wingman-Connect total training time is 5 hours, typically spread over three consecutive training 'blocks'(or days), plus 1-hour of booster training (one month later).
  Interventions: Behavioral: Wingman Connect
- Stress Management (Active Comparator): The control training condition will consist of a 2 hr. informational training that provides an overview of the human stress response system and strategies to manage stress. The training will be delivered through lecture format using PowerPoint, supplemented by brief videos and interactive discussion.
  Interventions: Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Wingman Connect — Wingman-Connect combines group and individual skill training. Group exercises build cohesion, belonging and shared purpose, and promote value of healthy unit, giving and receiving support. Individual skills promote the ability to thrive during transitions, manage stressors and meet career goals, and decrease barriers to utilizing organizational resources (family, health). The training has a total of 22 modules comprised of specific learning objectives and activities. Six months of text messages (1-2 per week) to reinforce and extend program concepts and skills.
  Arms: Wingman Connect
Behavioral: Stress Management — Stress management training reviews the basics of the hypothalamic-pituitary-adrenal axis stress-response system; common experiences of stress (physiological, cognitive, emotional); the impact of chronic stress on the brain and other domains of health; how exercise reduces harmful effects of stress; and relaxation techniques that have been shown to reduce stress and adverse effects of stress on health. Additional modules review the physiological stress response and effects of stress on health; introduces how cognition influences stress responses; common cognitive distortions/attributions are reviewed that affect stress including strategies to strengthen protective cognitive responses. Six months of text messages (1-2 per week) to reinforce and extend program concepts and skills.
  Arms: Stress Management

SUMMARY:
A study evaluating a training program to decrease risk for suicidal thoughts and behaviors among early career trainees in the United States Air Force.

DETAILED DESCRIPTION:
Relationship disruptions and social isolation are major precipitants for military suicides and a range of problems that impair functioning and reduce mission readiness. However, nearly all current military suicide prevention programming focuses on a narrow range of approaches for individuals already at high-risk (e.g., training to detect warning signs and refer for treatment services). This project addresses the need for universal prevention approaches to proactively strengthen protective factors across military populations, including strengthening social connectedness and skills to grow and sustain relationships across service.

The aims of this project are to (a) develop an intervention for early-career, enlisted United States Air Force personnel using an active training approach to strengthening social bonds, and (b) test the intervention (i.e., Wingman-Connect) using a randomized controlled trial design.

Wingman-Connect focuses on Airman-in-Training to build protective factors in: Kinship (healthy bonds); Guidance (support from mentors and mental health); Purpose (goals, sense of being valued and valuable); and Balance (self-care and support). Half of the training is focused on the class as a group to build belonging and shared purpose.

ELIGIBILITY:
Inclusion Criteria:

* Airmen-in-Training (AiT) in Technical Training classes in the 365 or 363 Training Squadrons of the 82 Training Wing (82 TRW)
* Eligible classes must be between 37-91 class days in length

Exclusion Criteria:

* Airmen from other countries receiving training in US
* Airmen who are not in their first year of enlistment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1485 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Wyman, PhD, Principal Investigator — University of Rochester Medical Center, Psychiatry Dept
Locations (1):
- Sheppard Air Force Base, Wichita Falls, Texas, United States

REFERENCES:
- [Background] Gibbons RD, Kupfer D, Frank E, Moore T, Beiser DG, Boudreaux ED. Development of a Computerized Adaptive Test Suicide Scale-The CAT-SS. J Clin Psychiatry. 2017 Nov/Dec;78(9):1376-1382. doi: 10.4088/JCP.16m10922. PMID 28493655
- [Background] Wyman PA, Brown CH, LoMurray M, Schmeelk-Cone K, Petrova M, Yu Q, Walsh E, Tu X, Wang W. An outcome evaluation of the Sources of Strength suicide prevention program delivered by adolescent peer leaders in high schools. Am J Public Health. 2010 Sep;100(9):1653-61. doi: 10.2105/AJPH.2009.190025. Epub 2010 Jul 15. PMID 20634440
- [Background] Petrova M, Wyman PA, Schmeelk-Cone K, Pisani AR. Positive-Themed Suicide Prevention Messages Delivered by Adolescent Peer Leaders: Proximal Impact on Classmates' Coping Attitudes and Perceptions of Adult Support. Suicide Life Threat Behav. 2015 Dec;45(6):651-63. doi: 10.1111/sltb.12156. Epub 2015 Feb 18. PMID 25692382
- [Background] Gibbons RD, Weiss DJ, Pilkonis PA, Frank E, Moore T, Kim JB, Kupfer DJ. Development of a computerized adaptive test for depression. Arch Gen Psychiatry. 2012 Nov;69(11):1104-12. doi: 10.1001/archgenpsychiatry.2012.14. PMID 23117634
- [Background] Herrell RK, Edens EN, Riviere LA, Thomas JL, Bliese PD, Hoge CW. Assessing functional impairment in a working military population: the Walter Reed functional impairment scale. Psychol Serv. 2014 Aug;11(3):254-64. doi: 10.1037/a0037347. PMID 25068298
- [Background] Williams, J, Brown, JM, Bray, RM, Anderson Goodell, EM, Olmsted, KR, Adler, AB. (2016) Unit Cohesion, Resilience, and Mental Health of Soldiers in Basic Combat Training, Military Psychology, 28:4, 241-250, DOI: 10.1037/mil0000120
- [Derived] Wyman PA, Pisani AR, Brown CH, Yates B, Morgan-DeVelder L, Schmeelk-Cone K, Gibbons RD, Caine ED, Petrova M, Neal-Walden T, Linkh DJ, Matteson A, Simonson J, Pflanz SE. Effect of the Wingman-Connect Upstream Suicide Prevention Program for Air Force Personnel in Training: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2022532. doi: 10.1001/jamanetworkopen.2020.22532. PMID 33084901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of classes was staggered over 16 months-Oct 2017 - Jan 2019-with classes matched. Clusters of class units within training squadron were formed over time as they became available, selected to maximize balance (e.g., AFSC), and randomized to one of two training conditions.
Groups:
- Stress Management: The control training condition will consist of a 2 hr. informational training that provides an overview of the human stress response system and strategies to manage stress.
  Stress Management: training reviews the basics of the hypothalamic-pituitary-adrenal axis stress-response system; common experiences of stress (physiological, cognitive, emotional); the impact of chronic stress on the brain and other domains of health; how exercise reduces harmful effects of stress; and relaxation techniques that have been shown to reduce stress and adverse effects of stress on health. Additional modules review the physiological stress response and effects of stress on health; how cognition influences stress responses; common cognitive distortions/attributions that affect stress including strategies to strengthen protective cognitive responses. Six months of text messages (1-2 per week) to reinforce and extend program concepts and skills.
Period: Overall Study
Arm/Group | Wingman Connect | Stress Management
Started | 748 | 737
Baseline Survey Completion | 746 | 735
1 Month Survey Completion | 697 | 694
6 Month Survey Completion | 629 | 618
Completed | 740 | 737
Not Completed | 8 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — no data provided | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stress Management: The control training condition will consist of a 2 hr. informational training that provides an overview of the human stress response system and strategies to manage stress.
  Stress Management: Stress management training reviews the basics of the hypothalamic-pituitary-adrenal axis stress-response system; common experiences of stress (physiological, cognitive, emotional); the impact of chronic stress on the brain and other domains of health; how exercise reduces harmful effects of stress; and relaxation techniques that have been shown to reduce stress and adverse effects of stress on health. Additional modules review the physiological stress response and effects of stress on health; introduces how cognition influences stress responses; common cognitive distortions/attributions are reviewed that affect stress including strategies to strengthen protective cognitive responses. Six months of text messages (1-2 per week) to reinforce and extend program concepts and skills.
- Total: Total of all reporting groups
Arm/Group | Wingman Connect | Stress Management | Total
Number analyzed (Participants) | 746 | 735 | 1481
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 746 | 735 | 1481
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.96 (3.255) | 20.87 (3.019) | 20.92 (3.140)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants in Wingman Connect and 4 participants in Stress Management did not report Sex in baseline survey
  Participants
    number analyzed (Participants) | 744 | 731 | 1475
    Female | 128 | 125 | 253
    Male | 616 | 606 | 1222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 154 | 291
  Not Hispanic or Latino | 608 | 581 | 1189
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — 47 in Wingman Connect and 46 in Stress Management reported 'Other' in race - these are included in the 'Not reported' category.
  Participants
    American Indian or Alaska Native | 6 | 5 | 11
    Asian | 31 | 31 | 62
    Native Hawaiian or Other Pacific Islander | 9 | 10 | 19
    Black or African American | 91 | 83 | 174
    White | 498 | 483 | 981
    More than one race | 59 | 72 | 131
    Unknown or Not Reported | 52 | 51 | 103
Educational Background [Count of Participants; unit: Participants]
  GED | 30 | 23 | 53
  High School Diploma | 597 | 571 | 1168
  Associates Degree | 72 | 87 | 159
  Bachelor's Degree or higher | 47 | 54 | 101
Military Component [Count of Participants; unit: Participants]
  Active Duty | 617 | 596 | 1213
  National Guard | 92 | 90 | 182
  Reserves | 37 | 49 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Computerized Adaptive Testing for Suicide Severity
Description: Participants will complete a computerized adaptive test for suicide severity. Participants will answer questions about their mental health. Participant scores will range from 0-100 with 100 indicating higher likelihood of current suicidal ideation and higher risk for suicide attempt.
Time Frame: 6 months
Population: Some participants completed the main survey, but not the computerized adaptive test section.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 577 | 571
units on a scale | 10.76 (13.87) | 12.12 (13.50)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .062, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = -0.13, 95% CI 2-sided [-.29 to .01]

2. Primary Outcome: Mean Computerized Adaptive Testing for Suicide Severity
Description: as for outcome 1
Time Frame: 1 month
Population: Some participants completed the main survey, but not the computerized adaptive test section.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 657 | 661
units on a scale | 11.05 (13.25) | 13.43 (13.94)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .001, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = -0.23, 95% CI 2-sided [-.39 to -.09]

3. Secondary Outcome: Mean Computerized Adaptive Testing for Depression
Description: Participants will complete a computerized adaptive test for depression. Participants will answer questions about their mental health. Participant scores will range from 0-100 with 100 indicating higher risk for clinical depression.
Time Frame: 6 months
Population: Some participants completed the main survey, but not the computerized adaptive test section.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 577 | 571
units on a scale | 13.36 (17.18) | 15.64 (15.21)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .027, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = -0.16, 95% CI 2-sided [-.34 to -.02]

4. Secondary Outcome: Computerized Adaptive Testing for Depression
Description: as for outcome 3
Time Frame: 1 month
Population: Some participants completed the main survey, but not the computerized adaptive test section.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 657 | 661
units on a scale | 15.42 (16.93) | 18.38 (16.87)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .002, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = -0.24, 95% CI 2-sided [-.41 to -.08]

5. Secondary Outcome: Mean Behavioral Occupational Performance Outcomes
Description: Participants will complete 5 yes/no questions about job performance, including if superior has expressed concerns about work performance, if Airman has received corrective training for substandard performance, received a negative counseling statement, received a Letter of Reprimand. The sum of affirmative responses will be calculated. Scores will range from 0-5 with 5 indicating greater work impairment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 629 | 618
units on a scale | 0.29 (0.93) | 0.28 (0.94)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .821, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = 0.01, 95% CI 2-sided [-.12 to .11]

6. Secondary Outcome: Mean Behavioral Occupational Performance Outcomes
Description: as for outcome 5
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 685 | 681
units on a scale | 0.17 (0.62) | 0.25 (0.73)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .024, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = -0.14, 95% CI 2-sided [-.31 to -.02]

7. Secondary Outcome: Mean Class Cohesion
Description: Participants will complete a 3-item scale on how well members of their class cooperate, can depend on each other and stand up for each other. Scores range from 0 to 4 with higher scores indicating higher class cohesion.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 687 | 698
units on a scale | 3.16 (0.72) | 3.05 (0.75)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .012, Mixed Models Analysis; Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = 0.18, 95% CI 2-sided [.04 to .29]

8. Secondary Outcome: Mean Number of Positive Connections to Classmates
Description: Participants will be asked to name up to 5 other students in their class who they respect and would choose to spend time with. Participants can name 0-5 classmates.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: classmates
Arm/Group | Wingman Connect | Stress Management
Number analyzed (Participants) | 687 | 698
classmates | 2.08 (1.61) | 1.83 (1.56)
Statistical Analysis 1: Comparison: Stress Management; Test type: Superiority; p = .010, Mixed Models Analysis — Model adjusts for class (random effect) and sex, age, race/ethnicity, and Air Force component; Effect size = 0.21, 95% CI 2-sided [.05 to .35]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Stress Management: The control training condition will consist of a 2 hr. informational training that provides an overview of the human stress response system and strategies to manage stress.
  Stress Management: Stress management training reviews the basics of the hypothalamic-pituitary-adrenal axis stress-response system; common experiences of stress (physiological, cognitive, emotional); the impact of chronic stress on the brain and other domains of health; how exercise reduces harmful effects of stress; and relaxation techniques that have been shown to reduce stress and adverse effects of stress on health. Additional modules review the physiological stress response and effects of stress on health; introduces how cognition influences stress responses; common cognitive distortions/attributions are reviewed that affect stress including strategies to strengthen protective cogn
Arm/Group | Wingman Connect | Stress Management
All-Cause Mortality (participants affected / at risk) | 0/748 | 0/737
Serious Adverse Events (participants affected / at risk) | 0/748 | 0/737
Other Adverse Events (participants affected / at risk) | 0/748 | 0/737

LIMITATIONS AND CAVEATS:
AiTs and training school leadership were not blinded to intervention condition. Second, outcomes relied on self-report. Third, trainers were research staff, and findings may not generalize to training by military personnel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04067401/Prot_SAP_000.pdf